CLINICAL TRIAL: NCT05627661
Title: Managing Multiple Seizure Types With Wearable Devices
Brief Title: Wearable Devices to Monitor Seizures in Autoimmune Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin H. Brinkmann, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 22-006702
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Autoimmune Epilepsy; Healthy
MeSH Terms: interventions — Biosensing Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autoimmune Epilepsy with Biosensors (Experimental): Subjects with suspected autoimmune epilepsy will wear biosensors on wrist or upper arm during the at home monitoring period.
  Interventions: Device: Biosensor
- Healthy Controls with Biosensors (Active Comparator): Neurologically normal adult healthy controls will wear biosensors on wrist or upper arm during the at home monitoring period.
  Interventions: Device: Biosensor

INTERVENTIONS:
Device: Biosensor — Noninvasive wearable biosensor device worn on the primary affected wrist or upper arm for as much time as is feasible for 7-10 days

SUMMARY:
The purpose of this research is to search for reproducible changes in a wide range of physical signals, including heart rate, muscle tone and activity and EEG before and at the onset of seizures in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with or suspected of having autoimmune epilepsy.
* Normal controls - cognitively normal subjects without epilepsy

Exclusion Criteria:

• Cognitive or psychiatric condition rendering patient unable to cooperate with data collection or manage and recharge smart watch and tablet computer devices. Presence of open or healing wounds near monitoring sites (infection risk).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Number of high-quality physiological signals | 10 days
  Total number of high-quality physiological signals recorded by biosensors
Number of Reproducible changes in physiological biosignals | 10 days
  Identification of reproducible changes in one or more physiological biosignals at onset of video and/or EEG-identified seizures

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Brinkmann, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials